CLINICAL TRIAL: NCT05769205
Title: Role of Multi Paramertic MRI and MRI Perfusion in Indetermint Ovarian Lesions by Using ORADS MRI
Brief Title: MRI in Ovarian Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Collaborators: principle investigator (Unknown)
Responsible Party: Principal Investigator, Maryam Farouk Mahmoud Sayed, Assiut university, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MRI in ovarian tumors
Record Dates: First submitted 2023-02-26; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Ovarian Neoplasms
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Intervention Model Description: females with ovarian masses
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- female with ovarian masses (Experimental): MRI with contrast according to the kidney function test of the patients
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MRI with contrast

SUMMARY:
Role of multi paramrtric MRI and MRI perfusion in indetermint ovarian lesions by using ORADS MRI

DETAILED DESCRIPTION:
Aim of study the purpose of this study is to investigate the capabilities of multi parametric MRI including DCE perfusion and DWI to discriminate between benign and malignant ovarian masses .

ELIGIBILITY:
Inclusion Criteria: females with ovarian masses

-

Exclusion Criteria:

* females with known benign ovarian masses

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Ovaries lesions
Enrollment: 25 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
MRI in ovarian tumors | 2 years
  Role of parametric MRI in determint ovarian lesions by using ORADS MRI

REFERENCES:
- [Background] Patel RK, Garg A, Dixit R, Gandhi G, Khurana N. The role of "penumbra sign" and diffusion-weighted imaging in adnexal masses: do they provide a clue in differentiating tubo-ovarian abscess from ovarian malignancy? Pol J Radiol. 2021 Dec 15;86:e661-e671. doi: 10.5114/pjr.2021.111986. eCollection 2021. PMID 35059059